CLINICAL TRIAL: NCT06707038
Title: Improving Access to Renal Transplantation for Underserved Black Communities
Acronym: AATAP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Federal funding was no longer viable
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Tampa General Hospital (Other)
Responsible Party: Principal Investigator, Daniela Ladner, Director, Northwestern University Transplant Outcomes Collaborative, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00223027; U01DK137258-01 (NIH)
Record Dates: First submitted 2024-11-21; First posted 2024-11-27 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant; ESRD (End Stage Renal Disease)
Keywords: Heath Services Research; Intervention
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Intervention Model Description: Investigators will use a 1:1 allocation ratio of randomization to intervention and control. Randomization will be stratified by sex (male, female) and age (divided into 2 categories). Participants will be assigned to a randomization group upon completing the eligibility screener and consent has been obtained, which will occur after the patient has attended the Roundtable visit and completed baseline questionnaires, but before their first visit with the center.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AATAP (intervention) Arm (Experimental): One clinic visit with all transplant providers, racially concordant care team, dedicated social worked. This will incorporate: Cultural congruency, trust, health literacy and psychological support. Questionnaires also to be administered
  Interventions: Behavioral: AATAP intervention
- Standard of Care (Control) Arm (No Intervention): Separate visits with nephologist, surgeons and social worker. This arm will follow common standard of care at the site. Questionnaires also to be administered

INTERVENTIONS:
Behavioral: AATAP intervention — AATAP is a program created to address the barriers that Black patients face when accessing transplantation. AATAP providers resources in cultural congruency, trust, psychosocial support, and health literacy to provide patients with the individualized support needed to access the kidney transplant waitlist
  Arms: AATAP (intervention) Arm

SUMMARY:
The goal of this clinical trial is to learn whether the African American Transplant Access Program can be successfully replicated at another large kidney transplant program. The main questions it aims to answer are:

Does the AATAP intervention increase the number of Black patients who are listed for kidney transplant? Does the AATAP intervention have an effect on Black patient self-efficacy and trust in care team?

Researchers will compare kidney transplant listing status after 12 months of patients in the AATAP intervention to usual care patients to see if the AATAP program increases the number of patients listed for transplant.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as Black or African American;
* 18 to 75 years of age
* have an eGFR < 20 or End Stage Renal Disease Diagnosis;
* screen positive for AATAP via the screener (for poor health literacy or poor medical adherence or psychosocial concerns);
* medically eligible to begin transplant evaluation process determined by transplant team

Exclusion Criteria:

* other racial groups
* participants who have previously received a transplant;
* pregnant women;
* participants who screen negative on the screener;
* children less than 18 years old

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-05-06 (Actual); Study Completion 2025-05-06 (Actual)

PRIMARY OUTCOMES:
Listing status for each Arm by month 12 | 12 months from time of enrollment
  Listing (active or inactive) status by month 12

SECONDARY OUTCOMES:
Quality of life using Patient-Reported Outcomes Measurement Information System (PROMIS) 1.2 Global Health Scale | at enrollment and at 12 months after enrollment
  Scoring/T-Score Metric: The T-score metric is standardized with a mean of 50 and a standard deviation (SD) of 10. This means a T-score of 50 represents the average score of the reference population, and each 10-point deviation represents one standard deviation above or below the mean.
  Minimum and Maximum Values: The T-score typically ranges from 20 to 80, though this can vary slightly depending on the specific population and scoring method used.
  Interpretation: Higher T-scores indicate better health outcomes, while lower T-scores indicate worse health outcomes.
Self-Efficacy in Kidney Dialysis Management using Perceived Kidney/Dialysis Self-Management Scale (PKDSMS) | at enrollment and at 12 months after enrollment
  Scoring: The PKDSMS uses an average score on a five-point Likert scale, where respondents rate their self-management abilities.
  Minimum and Maximum Values: The scale ranges from 1 to 5, with 1 indicating low self-efficacy and 5 indicating high self-efficacy.
  Interpretation: Higher scores indicate better self-management and higher confidence in managing kidney dialysis.
trust in care received by transplant team using Adapted Trust in Physicians Scale | at enrollment and at 12 months after enrollment
  Scoring: This scale typically uses a five-point Likert format, where respondents rate their level of agreement with various statements about their trust in their physicians. The response options range from "strongly disagree" to "strongly agree".
  Minimum and Maximum Values: The scale ranges from 1 to 5, with 1 indicating low trust and 5 indicating high trust.
  Interpretation: Higher scores indicate greater trust in the transplant team, while lower scores indicate less trust.

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Ladner, MD, MPH, FACS, FAST, Principal Investigator — Northwestern University
Locations (1):
- Tampa General Hospital, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No